CLINICAL TRIAL: NCT01880151
Title: NEw approacheS for The dIagnosis of AlzeiMer's diseAse Through neuroElectrical Changes in the Brain
Brief Title: Neuroelectrical Biomarkers for Alzheimer's Disease Stages
Acronym: ESTIMATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: C12-71; 2013-A00344-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Dementia; Prodromal; EEG; ERP; Biomarkers
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Electroencephalography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prodromal AD (Experimental): Presence of memory impairment Absence of impairment in activities of daily life EEG
  Interventions: Device: EEG
- Mild AD dementia (Experimental): Presence of memory impairment Presence of impairment in activities of daily life EEG
  Interventions: Device: EEG
- Healthy control group (Experimental): Absence of memory impairment Absence of impairment in activities of daily life Absence of known neurological conditions EEG
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — EEG recorded during a resting condition and during an episodic memory task condition
  Other Names: Electroencephalography; Electrical Geodesics Incorporated

SUMMARY:
Recent diagnostic criteria for Alzheimer's disease (AD) recognize an extended spectrum of AD stages as part of the disease, including a preclinical stage. This underscores the importance of early prognosis of AD when it is still possible to influence the course of the disorder. The investigators propose a comprehensive project which will target the data-driven modeling of the disease development. This goal will be achieved by creating and validating a battery of new sensitive biomarkers for clinical evaluation and prediction of AD in individuals. The AD-related brain changes will be assessed by noninvasive functional EEG measured during an episodic memory task in subjects at different stages of AD, as well as in healthy controls. The novel functional biomarkers will be extracted using a rigorous multistage selection procedure involving advanced methods for feature extraction, as well as statistics and classification for optimal selection. The ESTIMATE project will serve as a first step in an extensive array of research procedures which will enable the early clinical identification of Alzheimer's disease in elderly individuals who could then take advantage of preventive pharmaceutical therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age: 70-85 years old
* Presence of memory impairment
* Completed educational level: middle school
* Visual and auditory acuity: normal or corrected-to-normal

Exclusion Criteria:

* Monogenic AD
* Presence of a neurological disorder
* Stroke that has occurred in the last three months
* Prohibited medications
* Residence in skilled nursing facility
* Illiteracy, is unable to count or to read
* Claustrophobia

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-07-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Frequency band charactersitics of the electrophysiological brain response | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, PhD,MD,Prof, Principal Investigator — Institute of Memory and Alzheimer's Disease, Pitie-Salpetriere Hospital
Locations (1):
- Institute of Memory and Alzheimer's Disease, Pitie-Salpetriere Hospital, Paris, France